CLINICAL TRIAL: NCT04459065
Title: Evaluation of IRDye800CW-nimotuzumab in Lung Cancer Surgery
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Western Economic Diversification Canada (Other Government)
Responsible Party: Principal Investigator, Steven Bharadwaj, Thoracic surgeon, University of Saskatchewan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBIRD.20190430.Nimo800CW
Record Dates: First submitted 2020-06-22; First posted 2020-07-07 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: IRDye800CW; Nimotuzumab; Lung cancer; EGFR; Near infrared; Image guided surgery; Optical imaging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Single center, open-label, phase I/II image-guided surgery study to assess the image quality of IRDye800CW-nimotuzumab during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose intermediate time (Experimental): Participants will receive an i.v. infusion of 50 mg IRDye800CW-nimotuzumab. Participants will undergo lung cancer resection surgery 4-6 days after infusion. Vitals, blood sample and urine sample will be collected before infusion for a baseline. Blood and vitals will be taken post infusion. Blood and urine samples will be collected on the day of surgery. Participants will be followed up for any adverse event until day 30 post administration
  Interventions: Drug: IRDye800CW-nimotuzumab
- High dose intermediate time (Experimental): Participants will receive an i.v. infusion of 100 mg IRDye800CW-nimotuzumab. Participants will undergo lung cancer resection surgery 4-6 days after infusion. Vitals, blood sample and urine sample will be collected before infusion for a baseline. Blood and vitals will be taken post infusion. Blood and urine samples will be collected on the day of surgery. Participants will be followed up for any adverse event until day 30 post administration
  Interventions: Drug: IRDye800CW-nimotuzumab
- Optimal dose early time (Experimental): Participants will receive an i.v. infusion of 50 or 100 mg IRDye800CW-nimotuzumab (depending on results from cohorts 1 and 2). Participants will undergo lung cancer resection surgery 1-3 days after infusion. Vitals, blood sample and urine sample will be collected before infusion for a baseline. Blood and vitals will be taken post infusion. Blood and urine samples will be collected on the day of surgery. Participants will be followed up for any adverse event until day 30 post administration
  Interventions: Drug: IRDye800CW-nimotuzumab
- Optimal dose late time (Experimental): Participants will receive an i.v. infusion of 50 or 100 mg IRDye800CW-nimotuzumab (depending on cohorts 1 and 2). Participants will undergo lung cancer resection surgery 7+ days after infusion. Vitals, blood sample and urine sample will be collected before infusion for a baseline. Blood and vitals will be taken post infusion. Blood and urine samples will be collected on the day of surgery. Participants will be followed up for any adverse event until day 30 post administration
  Interventions: Drug: IRDye800CW-nimotuzumab

INTERVENTIONS:
Drug: IRDye800CW-nimotuzumab — 50 mg of IRDye800CW-nimotuzumab will be infused intravenously over a period of 30 minutes. Lung cancer resection surgery will be done at different time points post infusion

SUMMARY:
The purpose of this study is to determine the safety, optimal dose and imaging time of the investigational product, IRDye800CW-nimotuzumab for use as a near infrared imaging probe for image-guided surgery during lung cancer resection. IRDye800CW-nimotuzumab targets cancer cells over-expressing EGFR, allowing tumors to be visualized and may help surgeons better identify cancer during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Surgically resectable Stage I and II non-small cell lung cancer
* Able to give informed consent
* Age ≥ 18 and ≤ 80 years old
* Adequate cardiopulmonary reserve to undergo lung resection as determined by operating surgeon
* No prior history of malignancy
* No neoadjuvant therapy
* Karnofsky performance status of at least 70% or Eastern Cooperative Oncology Group (ECOG)/Zubrod level 0-2
* Hemoglobin (hgb) ≥ 90 g/L
* White blood cell count (WBC) > 3 x 109/L
* Platelet count (plt) ≥ 100 x 109/L
* Serum creatinine ≤ 1.5 times upper reference range

Exclusion Criteria:

* Received anti-EGFR antibody therapy (cetuximab, panitumumab, necitumumab) within 60 days prior to trial drug
* Pregnant or nursing
* Known history of hypersensitivities or allergic reactions to antibodies or NSO derived products
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* Subjects receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Optimal dose of IRDye800CW-nimotuzumab for image guided surgery. | up to 14 days
  To identify the dose with the highest tumor fluorescence and TBR.
Phase 2: Determine the optimal time for IRDye800CW-nimotuzumab infusion for image guided surgery. | up to 14 days
  To identify the imaging time with the highest tumor fluorescence and TBR.

SECONDARY OUTCOMES:
Determine primary tumor margins. | up to 14 days
  Determine the level of fluorescence that can discriminate between EGFR positive tumor tissue and normal tissue.
Identify EGFR positive lymph nodes. | up to 14 days
  Determine the level of fluorescence that can discriminate between EGFR positive lymph nodes and normal tissue.
Safety of IRDye800CW-nimotuzumab | up to 14 days
  a. Safety will be determined by recording the number of grade 2 or higher adverse events determined to be clinically significant, which are definitely, probably, or possibly related to IRDye800CW-nimotuzumab within 30 days of administration.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No